CLINICAL TRIAL: NCT03518879
Title: The ASTHMA-Educator: A Novel Algorithmic Software Tool to Help Manage Asthma
Brief Title: ASTHMA-Educator Mobile Application Manage Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013-2693
Record Dates: First submitted 2018-04-13; First posted 2018-05-08 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Asthma
Keywords: informatics; asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: This is a single-arm proof of concept study to evaluate the impact of the ASTHMA-Educator on process and clinical outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASTHMA-Educator arm (Experimental): The ASTHMA-Educator mobile application for patient-centered asthma education. The application is administered via on-site iPad (tablet).
  Interventions: Other: ASTHMA-Educator mobile application

INTERVENTIONS:
Other: ASTHMA-Educator mobile application — The on-site delivered ASTHMA-Educator mobile application.

SUMMARY:
Through this study, the investigators developed the ASTHMA-Educator mobile application, and evaluated its use among adult asthma patients at Montefiore.

DETAILED DESCRIPTION:
Through this study, the investigators developed the ASTHMA-Educator mobile application, and evaluated its use through 2 phases: 1) Phase 1 = process outcomes evaluation with 30 patients); and 2) Phase 2 (longitudinal clinical evaluation with 40 patients receiving the intervention at baseline, 2 months, 4 months, and 6 months). The study's primary outcome is asthma control.

ELIGIBILITY:
Inclusion Criteria: Adults (>18 years) with: (a) severe asthma (i.e. at least one asthma-related ED visit and/or hospitalization in the previous year); (b) access to a smartphone with short message service (SMS) capability; (c) English speaking; (d) able to give informed consent.

Exclusion Criteria: (a) use of oral corticosteroids in the 2 weeks prior to the baseline visit; (b) pregnancy; (c) severe psychiatric or cognitive problems that would prohibit an individual from understanding and completing the protocol; and (d) patients that previously received the ASTHMAXcel application.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline asthma control to 2, 4, and 6 months | Baseline, 2 months, 4 months, 6 months
  Asthma symptom burden as measured by the Asthma Control Test

SECONDARY OUTCOMES:
Change from baseline asthma knowledge to immediately post-intervention, 2 months, 4 months, and 6 months | Baseline, immediately post-intervention, 2 months, 4 months, 6 months
  Asthma knowledge as measured by the validated Asthma Knowledge Questionnaire
Patient satisfaction measured by the Client Satisfaction Questionnaire-8 | Immediately post-intervention at the baseline visit, 2 months, 4 months, 6 months
  Patient satisfaction measured by the Client Satisfaction Questionnaire-8
Time spent in using the mobile application | Immediately post-intervention at the baseline visit
  Time spent in using the mobile application
Asthma quality of life measured by the mini-Asthma Quality of Life Questionnaire (mini-AQLQ) | Baseline, 2 months, 4 months, 6 months
  Patients' asthma quality of life measured by the mini-Asthma Quality of Life Questionnaire (mini-AQLQ)
Asthma emergency department visits | Baseline, 2 months, 4 months, 6 months
  Asthma emergency department visits
Asthma hospitalizations | Baseline, 2 months, 4 months, 6 months
  Asthma hospitalizations
Asthma-related steroid courses | Baseline, 2 months, 4 months, 6 months
  Asthma-related steroid courses

CONTACTS AND LOCATIONS:
Overall Officials: Sunit Jariwala, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will share de-identified and aggregated study findings.